CLINICAL TRIAL: NCT03641118
Title: Assessment of Measures of Sarcopenia and Whole Body Physiology in Cancer Patients and Their Relationship to Surgical Outcome and Survival
Brief Title: Sarcopenia and Physiology Assessments in Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: University of Southampton (Other); Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: 16/SS/0188; 215694 (Other: IRAS project ID)
Record Dates: First submitted 2018-08-10; First posted 2018-08-21 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Upper Gastrointestinal Disorders; Lower Gastrointestinal Disorders; Hepatobiliary Cancer
Keywords: cancer; sarcopenia; surgery; chemotherapy
MeSH Terms: conditions — Gastrointestinal Diseases; Neoplasms; Sarcopenia | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Lower gastrointestinal cancer: All lower gastrointestinal neoplasms including rectal
  Interventions: Diagnostic Test: Cardiopulmonary exercise test
- Upper gastrointestinal cancer: All upper gastrointestinal neoplasms
  Interventions: Diagnostic Test: Cardiopulmonary exercise test
- Hepatobiliary cancers: All liver, pancreas, biliary cancer
  Interventions: Diagnostic Test: Cardiopulmonary exercise test

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary exercise test — The CPET test involves cycling on an exercise bike for 8-12 minutes. Starting with a very low resistance on the pedals the patient will pedal at 60 revolutions per minute. After 3 minutes of cycling, the resistance will gradually increase until the patient can no longer turn the pedals at the required speed. The test will be thoroughly explained to the patient beforehand and trained staff will make the experience as comfortable as possible. CPETs will be stopped early by the study researcher/doctor in the presence of any adverse events. Each CPET appointment will last approximately one hour.

SUMMARY:
Primary Aim:

To establish a reliable relationship between oxygen uptake (VO2) at estimated lactate threshold (AT) and CT-derived body composition measurments (e.g. muscle radiation attenuation), and to relate these to post-operative outcomes (i.e. post-operative complications or 1-year survival) in cohort of upper (UGI) and lower (LGI) gastrointestinal and hepatobiliary (HPB) cancer patients undergoing surgery +/- cancer therapies.

Rationale:Objectively measured reduction of muscle radiation attenuation (i.e. Computed Tomography (CT) measured indices of muscle wasting) coupled with reduced physical fitness (measured objectively using Cardiopulmonary Exercise Testing (CPET)) will result in worse post-operative surgical outcome and reduced survival.

Trial Design: Observational Sample size: See statistical analyses section for individual cohort power calculations Inclusion Criteria: Male or female patients, aged over 18 years old with UGI, LGI or HPB cancer undergoing surgery +/- cancer therapies; WHO performance status 0-2.

Exclusion Criteria: Patients will be excluded if they have surgery for benign disease, a diagnosis of inflammatory bowel disease, patients physically unable to perform a CPET on a cycle ergometer, patients having no surgery performed or interim emergency surgery, patients lacking complete in-hospital morbidity and survival data.

Primary Trial Endpoints: UGI patients - 2 year overall survival, LGI and HPB patients - post-operative complications (Calvien-Dindo and Composite Endpoint in pancreaticoduodenectomy)

DETAILED DESCRIPTION:
Study overview and background

We hypothesise that an objectively measured reduction in muscle radiation attenuation (i.e. Computed Tomography (CT) measured indices of muscle wasting and/or sarcopenia) coupled with reduced physical fitness (measured objectively using Cardiopulmonary Exercise Testing (CPET)) will result in worse post-operative surgical outcome and reduced survival in patients going straight to surgery or having cancer therapies.

An analyses of prospectively collected clinical data from routine clinical practice in a cohort of upper and lower gastrointestinal and hepatobiliary (liver, pancreas and biliary tree) cancer patients will be undertaken. These patients may undergo neoadjuvant (before surgery) cancer therapies before undergoing surgery.

We aim to interrogate prospectively collected objectively measures of radiological markers of muscle wasting and body composition, as well as objectively measured markers of physical fitness in 3 cohorts: upper and lower gastrointestinal and hepatobiliary (liver, pancreas and biliary tree) cancer patients and to explore if body composition is related with physical fitness. In addition, body composition and physical fitness will be related to post-operative outcomes and survival. These data will be readily available as they are collected as part of routine clinical care at University Hospital Southampton NHS Foundation Trust. Our hospital performs a large number of major cancer operations in these 3 cancer patient groups. These patients already undergo accurate radiological cancer staging and sometimes re-staging (after cancer therapies) and also a CPET as part of their pre-operative pathway. As part of their enhanced recovery pathway, which is now well embedded into routine clinical care, post-operative surgical outcomes, cancer outcomes and survival are routinely collected.

METHODOLOGY

Patients will be identified from prospectively maintained enhanced recovery databases. All patients will be having surgery at University Hospital Southampton where all upper and lower gastrointestinal and hepatobiliary (liver, pancreas and biliary tree) cancer teams maintain well validated enhanced recovery databases with patient and cancer specific demographics, operative records, histopathological, cancer specific and post-operative outcomes. These databases are maintained to a high level due to their usage in national cancer audits. All patients will undergo a staging CT (as part of routine care), this will be used to measure radiological markers of sarcopenia and body composition in the research setting. No additional radiological scanning sequences, contrast or scanner time is required here. In addition all patients will also undergo a CPET (also as part of routine care), this will be used to objectively measure markers of pre-operative physical fitness. The CPET protocol is defined in Appendix 1 of the trial protocol. All variables measured by CT and CPET that will be collected are outlined in Appendix 2 of the trial protocol.

Following staging investigations patients may undergo neoadjuvant cancer treatments. Re-staging radiological investigations will be performed as part of standard care in all 3 cohorts. All patients will undergo major cancer specific surgical procedures. Following surgery routinely collected clinically relevant observational data will be used to define post-operative outcomes. These data will relate to hospital length of stay, the level intensive or high dependency care required following surgery, post-operative morbidity (Postoperative Morbidity Survey - POMS and Clavine-Dindo Score) and survival. Most of this information can be accessed from prospectively maintained enhanced recovery databases; however patient notes and electronic patient records are acceptable alternatives. All of these data are already collected as part of routine care and not additional resources for data collection will be required. Appendix 2 shows the minimum dataset that will be collected. Survival at 2 years will be collected for all patients.

All patients will be given a patient information sheet and formally consented to ask for their permission for these data to be used for research purposes.

Contraindications to CPET based on ACCP/ATS Guidelines are summarised in the American Journal of Respiratory and Critical Care Medicine 2003; 167: 211-77.

Please see also for further information:

http://www.thoracic.org/statements/resources/pfet/cardioexercise.pdf http://www.pcpet.co.uk/Links

HYPOTHESIS

We hypothesise that an objectively measured reduction of muscle radiation attenuation (i.e. Computed Tomography (CT) measured indices of myosteatosis) is related to reduced physical fitness (measured objectively using Cardiopulmonary Exercise Testing (CPET)) and both will result in worse operative or cancer progression related outcome and reduced survival.

Specifically we aim to interrogate the relationship between oxygen uptake (Vo2) at estimated lactate threshold (LT) and muscle radiation attenuation and post-operative outcomes (i.e. post-operative complications - LGI and HPB cohorts and 2-year survival - UGI cohort) in patients undergoing surgery +/- neoadjuvant cancer therapies.

DATA ANALYSES - CT-scan analysis and data transfer

Abdominal CT-scans will be analysed in anonymized format by one blinded independent researcher trained in radiologic anatomy and body composition analysis. These analyses will be done at the University of Maastricht by Prof Steven Olde Damnik. A single fully anonymised CT image (as described hereunder) will be sent to Prof Olde Damnik using encrypted software using encrypted and password protected hardware (NHS purchased Safe Stick). No other data will be sent to Maastricht. This image will be processed and data relating to variables below will be sent back to the PI. All other data analyses will be done by the PI at University Hospitals Southampton. All data will be stored, processed and analysed on secure NHS computers on NHS encrypted and password-protected servers used by the Critical Care Research Team.

A single slice of each patient's CT-scan will be selected at the level of the third lumbar vertebra (L3). CT-scans with large radiation artefacts or with missing parts of muscle tissue on the ventral, dorsal, or both lateral edges of the scan will be excluded. Muscles included into the analysis are the internal and external obliques, transversus abdominus, rectus abdominus, psoas, quadratus lumborum, and erector spinae muscles. CT-scans will be analysed using sliceOmatic 5.0 (TomoVision, Magog, Canada) software for Microsoft Windows®. Using predefined Hounsfield unit (HU) ranges, the total cross-sectional area (cm2) of skeletal muscle tissue ( 29 to 150 HU), visceral adipose tissue (VAT; -150 to 50 HU), subcutaneous adipose tissue (SAT; 190 to 30 HU), and intermuscular adipose tissue (IMAT; 190 to 30 HU) will be determined. In addition, the radiation attenuation for skeletal muscle will be assessed by calculating the average HU value of the total muscle area within the specified range of -29 to 150 HU (i.e. this is calculated from the muscle tissue only excluding the IMAT). The total areas of skeletal muscle, VAT and SAT will be corrected for stature to calculate the L3-muscle index, L3-VAT index, and L3-SAT index in cm2/m2, providing good estimates of total body skeletal muscle, VAT, and SAT mass.

Cardiopulmonary Exercise Tests (CPET)

The CPET test involves cycling on an exercise bike for 8-12 minutes. Starting with a very low resistance on the pedals the patient will pedal at 60 revolutions per minute. After 3 minutes of cycling, the resistance will gradually increase until the patient can no longer turn the pedals at the required speed. The test will be thoroughly explained to the patient beforehand and trained staff will make the experience as comfortable as possible. CPETs will be stopped early by the study researcher/doctor in the presence of any adverse events. Each CPET appointment will last approximately one hour.

CPETs carry a small risk (1:10,000) of exercise induced myocardial infarction or dysrhythmia. Patients are continuously monitored using a 12 lead electrocardiograph (ECG) during all tests and recovery. The CPET test will entail the patient becoming slightly hot or maybe sweaty, and appropriate clothing should be worn. The patient's heart will be monitored by an electrocardiogram. The patient will wear a soft rubber mask in order to continuously sample expired air with an online breath by breath gas analyzer. This may cause some mild claustrophobia. Full detail of the CPET procedure is given in appendix 1. Physiologists with experience in analysis of exercise tests will analyse all of the exercise data. Patients will be anonymised and the physiologist performing the data analysis will be blinded to the sarcopenia measurements and the outcome data. All data will be stored, processed and analysed on secure NHS computers on NHS encrypted and password-protected servers used by the Critical Care Research Team.

STATISTICAL METHODOLOGY

For all CT body composition measurements, sex-specific cut-offs will be determined at the median. The main parameter will be muscle radiation attenuation, as this parameter was found to have the most effect on post-operative complications in our previous study. Data will be analysed using IBM SPSS 23 for Microsoft Windows®. Differences in patient characteristics will be analysed using the independent T-test or Pearson chi-square test. The Pearson chi-square test will be used to assess the difference in post-operative complications or survival; for patients with low vs. high muscle radiation attenuation and other body composition measurements. For correlations, Pearson's correlation coefficient (rp) will be used. A p-value of <0.05 was considered significant.

Power analysis

HPB cohort

The sample sizes calculation for this study were determined using our previous results in a Dutch pancreatic cancer patient cohort. In this study, the occurrence of the CEP was compared between patients with HPB cancer and a low muscle radiation versus high muscle radiation attenuation. We found a significantly higher CEP occurrence in the low muscle radiation group (p=0.027). Using this population (n=184) we calculated an effect size (w) of 0.331. Using this effect size we conducted a power analysis for the HPB cohort with a power of 0.80 and an α of 0.05 considered as significant which resulted in a total sample size of 72 patients.

Upper gastrointestinal cancer cohort

The sample size calculation for this study was based on a study by Yip et al. We are planning a study with one control per experimental subject, an accrual interval of 9 months, and additional overall survival follow-up after the accrual interval of 24 months. Prior data indicate that the median survival time on the control treatment is 25.6 months. If the true median survival times on the control and experimental treatments are 25.6 and 55 months, respectively, we will need to study 138 patients to be able to reject the null hypothesis that the experimental and control survival curves are equal with probability (power) 0.800. The Type I error probability associated with this test of this null hypothesis is 0.05.

Lower gastrointestinal cancer cohort

The sample size calculation for this study was based on a study by Lieffers et al. Prior data indicate a 24% post-operative complication rate in the sarcopenia group as opposed to a 13% complication rate in the non-sarcopenia group (OR 0.460). We will need to study 404 patients with probability (power) 0.800. The Type I error probability associated with this test of this null hypothesis is 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* aged over 18 years old
* undergoing surgery and/or cancer therapies
* WHO performance status 0-2.

Exclusion Criteria:

* benign disease
* a diagnosis of inflammatory bowel disease
* patients physically unable to perform a CPET on a cycle ergometer
* patients having no surgery performed or interim emergency surgery
* patients lacking complete in-hospital morbidity and survival data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Upper gastrointestinal cancer, lower gastrointestinal cancer or hepatobiliary cancers
Sampling Method: Probability Sample
Enrollment: 639 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle radiation attenuation at L3 | up to 4 week before surgery
  muscle radiation attenuation using CT L3 image slice using Slico-matic software

SECONDARY OUTCOMES:
Surgical morbidity | throughout study completion whilst patient is in hospital, up to 6 months
  Clavien-dindo complication
Survival | at 1 year after surgery
  1-year survival
oxygen uptake at lactate threshold | up to 4 weeks before surgery
  Cardiopulmonary exercise testing

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm West, PhD, Principal Investigator — University Hospitals Southampton NHS Foundation Trust
Locations (1):
- University Hospitals Southampton, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual patient data to be shared